CLINICAL TRIAL: NCT02175615
Title: PHARMACOLOGICAL PREDICTORS OF SUCCESSFUL CYCLOSPORINE ACUTE GRAFT VERSUS HOST DISEASE PROPHYLAXIS IN CHILDREN UNDERGOING HAEMATOPOIETIC STEM CELL TRANSPLANT
Brief Title: Pharmacological Predictors of Successful Cyclosporine Acute GVHD Prophylaxis in Children Undergoing HSCT
Status: Completed | Type: Observational
Sponsor: Lee Dupuis (Other)
Collaborators: C17 Council (Other)
Responsible Party: Sponsor-Investigator, Lee Dupuis, Dr. Lee Dupuis, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: CSA Cyclosporine PK Study
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Acute-graft-versus-host Disease
Keywords: CYCLOSPORINE; ACUTE GRAFT VERSUS HOST DISEASE; PROPHYLAXIS; CHILDREN; HAEMATOPOIETIC STEM CELL TRANSPLANT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The specific objectives of this study are:

Primary:

1)To determine the relationship between cyclosporine AUC achieved prior to engraftment and severe aGVHD (grade III and IV)

Secondary:

1. To determine the relationship between individual concentration-time points achieved prior to engraftment and severe aGVHD (grade III and IV)
2. To validate the previously developed LSS to determine cyclosporine AUC after IV administration at steady state and
3. To describe the relationship between cyclosporine AUC and individual concentration-time points achieved prior to engraftment and other HSCT outcomes (clinically significant aGVHD (grade II to IV), hypertension, engraftment failure, relapse

ELIGIBILITY:
Inclusion Criteria:

* less than 18 years of age
* undergoing allogeneic myeloablative HSCT at one of the participating centres and
* scheduled to receive cyclosporine for aGVHD prophylaxis
* minimum patient weight:
* 6.4kg if < 6 months old or 7.2kg if > 6 months old

All patients or guardians will provide informed consent or assent as appropriate. Initial contact will be made by a member of the patient's current care team. Consent will be obtained by a co-investigator or the CTSU personnel.

Exclusion Criteria:

-receipt of voriconazole or posaconazole within 14 days of the first cyclosporine dose or at any time until engraftment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ALLOGENEIC Hematopoietic stem cell transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Relationship between CSA area-under-the-curve (AUC) prior to ENGRAFTMENT and severe aGVHD | Weekly for 7 weeks or until engraftment and for 100 days after HSCT
  1)To determine the relationship between cyclosporine AUC achieved prior to engraftment and severe aGVHD (grade III and IV)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dupuis, PhD, Principal Investigator — SickKids Research Institute
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Dupuis LL, Seto W, Teuffel O, Gibson P, Schultz KR, Doyle JD, Gassas A, Egeler RM, Sung L, Schechter T. Prediction of area under the cyclosporine concentration versus time curve in children undergoing hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2013 Mar;19(3):418-23. doi: 10.1016/j.bbmt.2012.10.031. Epub 2012 Nov 2. PMID 23128321